CLINICAL TRIAL: NCT04569513
Title: The Analysis of Thyroidectomy and Parathyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201906051RINA
Record Dates: First submitted 2020-05-11; First posted 2020-09-30 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Thyroid Diseases; Parathyroid Diseases
Keywords: surgery; ablation; minimal invasive surgery
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases | interventions — Thyroid (USP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Thyroid and parathyroid disease — To analyze surgery or not, different surgical methods, timing of surgery, and alternative managements for patients of thyroid or parathyroid disease.

SUMMARY:
To analyze surgery or not, different surgical methods, timing of surgery, and alternative managements for patients of thyroid or parathyroid disease.

DETAILED DESCRIPTION:
Utilizing our institutional database, tissue bank, and electronic medical charts to surgery or not, different surgical methods, timing of surgery, and alternative managements for patients of thyroid or parathyroid disease.

ELIGIBILITY:
Inclusion Criteria:

* age more than 20 years
* thyroid or parathyroid disorder
* willing to receive management at National Taiwan University Hospital (NTUH)

Exclusion Criteria:

* age less than 20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of thyroid or parathyroid disorder at National Taiwan University Hospital (NTUH).
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2021-06-10 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 month
  Death or live
Progression | 1 month
  Recurrence or metastasis

SECONDARY OUTCOMES:
Tumor growth | 1 cm/month
  Size variation of tumor
Life quality | 1 year
  Cosmetic and symptoms, using short-form (SF)-36 and patient satisfaction scale (as tumor volume reduction rate, satisfy as >50%)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hsun Wu, MDPhD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- Ting-Chun Kuo, Taipei, Taiwan